CLINICAL TRIAL: NCT00454389
Title: A Randomized, Prospective, Active Controlled, Study of the Epi-Rad90™ Ophthalmic System for the Treatment of Subfoveal Choroidal Neovascularization Associated With Wet Age-Related Macular Degeneration
Brief Title: A Study of Strontium90 Beta Radiation With Lucentis to Treat Age-Related Macular Degeneration
Acronym: CABERNET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeoVista (Industry)
Responsible Party: NeoVista, Inc./Jeffrey A. Nau, MMS, Director of Clinical Affairs, NeoVista, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVI-114
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Macular Degeneration
Keywords: Macular; Degeneration; AMD; Wet Age-Related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Epi-Rad90™ Ophthalmic System procedure + Lucentis
  Interventions: Device: Epi-Rad90™ Ophthalmic System
- B (Active Comparator): Lucentis only
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Device: Epi-Rad90™ Ophthalmic System — A single procedure using the Epi-Rad90™ Ophthalmic System plus 2 injections of Lucentis administered 1 month apart
  Arms: A
Drug: ranibizumab — Lucentis injection administered monthly for the first 3 injections followed by quarterly injections
  Other Names: Lucentis
  Arms: B

SUMMARY:
The objective of the CABERNET Trial is to evaluate the safety and efficacy of focal delivery of radiation for the treatment of subfoveal choroidal neovascularization (CNV) associated with wet age-related macular degeneration (AMD). The Epi-Rad90™ Ophthalmic System treats neovascularization of retinal tissue by means of a focal, directional delivery of radiation to the target tissues in the retina. Using standard vitreoretinal surgical techniques, the sealed radiation source is placed temporarily over the retinal lesion by means of a handheld medical device.

DETAILED DESCRIPTION:
Therapeutic advances in the arena of neovascular age-related macular degeneration (AMD) have provided multiple treatment options for the disease. Radiotherapy has been studied in multiple clinical trials in the past with many studies showing a therapeutic benefit. Treatment with radiotherapy and anti-VEGF compounds is a promising approach to treating AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have predominantly classic, minimally classic, or occult with no classic lesions, as determined by the Investigator, secondary to AMD, with a total lesion size (including blood, scarring, and neovascularization) of < 12 total disc areas (21.24 mm2), and a GLD ≤5.4 mm
* Subjects must be age 50 or older

Exclusion Criteria:

* Subjects with prior or concurrent subfoveal CNV therapy including thermal laser photocoagulation (with or without photographic evidence), photodynamic therapy, injections with Macugen®, intravitreal or subretinal steroids, transpupillary thermotherapy (TTT), and systemic anti-angiogenic or intravitreal anti-angiogenic agents in study eye. (Note: This includes subjects with no known history, but with photographic evidence of prior therapy)
* Subjects who underwent previous radiation therapy to the eye, head or neck
* Subjects that have been previously diagnosed or have retinal findings consistent with Type 1 or Type 2 Diabetes Mellitus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects losing fewer than 15 letters of best corrected visual acuity score at 12 months compared to baseline. Gain of 15 more letters of best correct visual acuity score compared to baseline | 12 months

SECONDARY OUTCOMES:
No loss in ETDRS letters | 12 months
Change in total lesion size and CNV size by fluorescein angiography | 12 months
Number of rescue injections of Lucentis. | 12 months
Mean change in ETDRS visual acuity | 12 months
Incidence and severity of adverse events and ocular adverse events. Incidence of cataract changes. Incidents of radiation induced toxicity. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pravin Dugel, MD, Principal Investigator — Retinal Consultants of Arizona; Jeffrey A Nau, MMS, Study Director — NeoVista, Inc.
Locations (32):
- United States (23):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina Center, PC, Tucson, Arizona
  - Retina-Vitreous Associates Medical, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - UCSF Koret Vision Center, San Francisco, California
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Retina Institute of Hawaii, Honolulu, Hawaii
  - Paducah Retinal Center, Paducah, Kentucky
  - New England Eye Center-Tufts University, Boston, Massachusetts
  - Associated Retinal Consultants / William Beaumont Hospital, Royal Oak, Michigan
  - Eye Foundation of Kansas City, Kansas City, Missouri
  - Charlotte Eye Ear Nose & Throat Associates, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Research Unit of Wills Eye Hospital, Philadelphia, Pennsylvania
  - Tennessee Retina, Nashville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina & Uveitis Consultants of Texas, San Antonio, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- Augenklinik Graz, Graz, Austria
- Germany (2):
  - Klinik und Poliklinik für Augenheilkunde der Universität Leipzig AöR, Leipzig
  - Universitätsklinik und polyklinik für Augenkranke, Würzburg
- Institute of Clinical Science, Ophthalmic Research Centre, Royal Victoria Hospital, Belfast, Ireland
- Sourasky Medical Center, Tel Aviv, Israel
- Oftalmo Salud Eye Institute, Lima, Peru
- Institutio de Microcirugia Ocular-Barcelona, Barcelona, Spain
- University of Geneva, Geneva, Switzerland
- Kings College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Evans JR, Igwe C, Jackson TL, Chong V. Radiotherapy for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 Aug 26;8(8):CD004004. doi: 10.1002/14651858.CD004004.pub4. PMID 32844399